CLINICAL TRIAL: NCT04903509
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Subcutaneous Doses of BI 1820237 Alone (Trial Parts 1+2) or Together With a Low Dose of Liraglutide (Trial Part 3) in Otherwise Healthy Male Subjects With Overweight/Obesity (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Men With Overweight to Test How Well Different Doses of BI 1820237 Are Tolerated When Given as an Injection Alone or in Combination With Liraglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1458-0001; 2021-000327-13 (EudraCT Number)
Record Dates: First submitted 2021-05-25; First posted 2021-05-26 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — Liraglutide; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Masking Description: Within the central electrocardiogram (ECG) lab, the staff involved with interval measurements will be blinded with respect to the treatment and also with regard to the recording date and time as well as planned time points of the ECGs. The interval measurements for a given subject will be performed in a random and blinded sequence by a single technician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BI 1820237 (Experimental): Part 1 and part 2 of the trial.
  Interventions: Drug: BI 1820237; Drug: Paracetamol-ratiopharm®
- Placebo (Placebo Comparator): Part 1 and part 2 of the trial.
  Interventions: Drug: Placebo; Drug: Paracetamol-ratiopharm®
- BI 1820237 + liraglutide (Experimental): Part 3 of the trial.
  Interventions: Drug: BI 1820237; Drug: Saxenda®; Drug: Paracetamol-ratiopharm®
- Placebo + liraglutide (Placebo Comparator): Part 3 of the trial.
  Interventions: Drug: Placebo; Drug: Saxenda®; Drug: Paracetamol-ratiopharm®

INTERVENTIONS:
Drug: BI 1820237 — BI 1820237
  Arms: BI 1820237; BI 1820237 + liraglutide
Drug: Placebo — Placebo
  Arms: Placebo; Placebo + liraglutide
Drug: Saxenda® — Saxenda®
  Other Names: Liraglutide
  Arms: BI 1820237 + liraglutide; Placebo + liraglutide
Drug: Paracetamol-ratiopharm® — Paracetamol-ratiopharm®
  Other Names: Paracetamol

SUMMARY:
The main objective of this trial is to investigate safety, tolerability and pharmacokinetics (PK) and pharmacodynamics (PD) of BI 1820237 alone or together with a single low dose of liraglutide in male subjects with overweight/obesity (otherwise healthy) following subcutaneous administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with overweight/obesity (otherwise healthy) according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12 lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 25.0 to 34.9 kg/m2 (inclusive). Overweight should be due to excess adipose tissue, as judged by the investigator
* Body weight greater than or equal to 70 kg
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medications except appendectomy or simple hernia repair
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related adverse events | up to 48 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 38 days
Maximum measured concentration of the analyte in plasma (Cmax) | up to 38 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. Studies in products where Boehringer Ingelheim is not the license holder;
  2. Studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com